CLINICAL TRIAL: NCT01760889
Title: A Phase 3 Multicenter, Randomized, Double-blind, Parallel-group, Placebo-controlled, 26-week, Dose-optimization Study to Evaluate the Efficacy, Safety, and Tolerability of SPD489 Low Dose Range (40mg, 80mg, 100mg) and High Dose Range (120mg, 140mg, 160mg) as Adjunctive Treatment to Established Maintenance Doses of Antipsychotic Medications on Negative Symptoms in Clinically Stable Adults Who Have Persistent Predominant Negative Symptoms of Schizophrenia
Brief Title: SPD489 Low Dose and High Dose Ranges When Added to Stable Doses of Antipsychotic Medications in Clinically Stable Adults With Negative Symptoms of Schizophrenia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was discontinued due to non-safety related business prioritization decisions. No subjects were randomized
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPD489-335; 2012-003919-57 (EudraCT Number)
Record Dates: First submitted 2013-01-02; First posted 2013-01-04 (Estimated); Results first posted 2014-05-29 (Estimated); Last update posted 2021-06-22 (Actual); Status verified 2021-05

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Lisdexamfetamine Dimesylate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- SPD489 Low Dose Range (Experimental)
  Interventions: Drug: SPD489 low dose range (40mg, 80mg, and 100mg)
- SPD489 High Dose Range (Experimental)
  Interventions: Drug: SPD489 high dose range (120mg, 140mg and 160mg)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SPD489 low dose range (40mg, 80mg, and 100mg) — Capsule, dose titration,
  * 40 mg capsule once-daily for 1 week; then
  * 80 mg capsule once-daily for 4 weeks; then,
  * 100 mg capsule once-daily (if unable to tolerate 100 mg dose between weeks 5 to 6, then dose to be decreased to 80 mg once-daily for the remaining 21 weeks;
  * if able to tolerate 100 mg dose then will continue on 100 mg capsule once-daily for 21 weeks
  Other Names: lisdexamfetamine dimesylate, LDX, Vyvanse
  Arms: SPD489 Low Dose Range
Drug: SPD489 high dose range (120mg, 140mg and 160mg) — Capsule, dose titration,
  * 40 mg capsule once-daily for 1 week; then
  * 80 mg capsule once daily for 1 week; then
  * 120 mg capsule once-daily for 1 week, then,
  * 140 mg capsule once-daily for 2 weeks, then
  * 160 mg once capsule once-daily (if unable to tolerate 160 mg dose between weeks 5 to 6, then dose to be decreased to 140 mg once-daily for the remaining 21 weeks;
  * if able to tolerate 160 mg dose then will continue on 160 mg capsule once-daily for 21 weeks
  Other Names: lisdexamfetamine dimesylate, LDX, Vyvanse
  Arms: SPD489 High Dose Range
Drug: Placebo — One capsule a day for 26 weeks
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to determine whether SPD489 low dose range (40, 80, or 100mg) and high dose range (120, 140, or 160mg) are effective in the treatment of Negative Symptoms.

ELIGIBILITY:
Inclusion Criteria:

* - 18 to 65 years of age
* Has a reliable informant (eg, family member, social worker, caseworker, or nurse that spends >4 hours/week with the subject)
* Fixed home/place of residence and can be reached by telephone
* On a stable dose of antipsychotic medications
* Able to swallow capsules

Exclusion Criteria:

* Taking lithium, carbamazepine, lamotrigine, gabapentin, cholinesterase inhibitors, modafinil, or other stimulants such as methylphenidate and other amphetamine products
* Treated with clozapine in past 30 days
* Lifetime history of stimulant, cocaine, or amphetamine abuse or dependence
* History of seizures (other than infantile febrile seizures), any tic disorder, or current diagnosis and/or a known family history of Tourette's Disorder, serious neurological disease, history of significant head trauma, dementia, cerebrovascular disease, Parkinson's disease, or intracranial lesions
* Uncontrolled hypertension
* History of thyroid disorder that has not been stabilized on thyroid medication
* Glaucoma
* Pregnant or nursing
* Subject has received an investigational product or participated in a clinical study within 30 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-02-01 (Actual); Primary Completion 2013-04-01 (Actual); Study Completion 2013-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (4):
- United States (4):
  - Galiz Research, Miami Springs, Florida
  - Psychiatric Care and Research Center, O'Fallon, Missouri
  - St. Charles Psychiatric Associates, Saint Charles, Missouri
  - CRI Lifetree, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study was discontinued due to non-safety related business prioritization decisions. No subjects were randomized
Groups:
- SPD489 Low Dose Range: SPD489 low dose range (40mg, 80mg, and 100mg): Capsule, dose titration, • 40 mg capsule once-daily for 1 week; then • 80 mg capsule once-daily for 4 weeks; then, • 100 mg capsule once-daily (if unable to tolerate 100 mg dose between weeks 5 to 6, then dose to be decreased to 80 mg once-daily for the remaining 21 weeks; • if able to tolerate 100 mg dose then will continue on 100 mg capsule once-daily for 21 weeks
- SPD489 High Dose Range: SPD489 high dose range (120mg, 140mg and 160mg): Capsule, dose titration, • 40 mg capsule once-daily for 1 week; then • 80 mg capsule once daily for 1 week; then • 120 mg capsule once-daily for 1 week, then, • 140 mg capsule once-daily for 2 weeks, then • 160 mg once capsule once-daily (if unable to tolerate 160 mg dose between weeks 5 to 6, then dose to be decreased to 140 mg once-daily for the remaining 21 weeks; • if able to tolerate 160 mg dose then will continue on 160 mg capsule once-daily for 21 weeks
Period: Overall Study
Arm/Group | SPD489 Low Dose Range | SPD489 High Dose Range | Placebo
Started | 0 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Study was discontinued due to non-safety related business prioritization decisions. No subjects were randomized
Groups:
- Total: Total of all reporting groups
Arm/Group | SPD489 Low Dose Range | SPD489 High Dose Range | Placebo | Total
Number analyzed (Participants) | 0 | 0 | 0 | 0
Age, Categorical
Sex: Female, Male
Region of Enrollment

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Negative Symptom Assessment (NSA-16) Total Score at 26 Weeks
Time Frame: Baseline and 26 weeks
Population: Study was discontinued due to non-safety related business prioritization decisions. No subjects were randomized
Arm/Group | SPD489 Low Dose Range | SPD489 High Dose Range | Placebo
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Change From Baseline in the Personal and Social Performance (PSP) Scale Score at 26 Weeks
Time Frame: Baseline and 26 weeks
Population: Study was discontinued due to non-safety related business prioritization decisions. No subjects were randomized
Arm/Group | SPD489 Low Dose Range | SPD489 High Dose Range | Placebo
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Change From Baseline in Simpson Angus Scale (SAS) Total Score at 26 Weeks
Time Frame: Baseline and 26 weeks
Population: Study was discontinued due to non-safety related business prioritization decisions. No subjects were randomized
Arm/Group | SPD489 Low Dose Range | SPD489 High Dose Range | Placebo
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Change From Baseline in Barnes Akathisia Scale (BAS) Total Score at 26 Weeks
Time Frame: Baseline and 26 weeks
Population: Study was discontinued due to non-safety related business prioritization decisions. No subjects were randomized
Arm/Group | SPD489 Low Dose Range | SPD489 High Dose Range | Placebo
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Change From Baseline in the Abnormal Involuntary Movement Scale (AIMS) at 26 Weeks
Time Frame: Baseline and 26 weeks
Population: Study was discontinued due to non-safety related business prioritization decisions. No subjects were randomized
Arm/Group | SPD489 Low Dose Range | SPD489 High Dose Range | Placebo
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Scores at 26 Weeks
Time Frame: Baseline and 26 weeks
Population: Study was discontinued due to non-safety related business prioritization decisions. No subjects were randomized
Arm/Group | SPD489 Low Dose Range | SPD489 High Dose Range | Placebo
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Change From Baseline in Cognitive Test Battery (CogState Battery) Score at 26 Weeks
Time Frame: Baseline and 26 weeks
Population: Study was discontinued due to non-safety related business prioritization decisions. No subjects were randomized
Arm/Group | SPD489 Low Dose Range | SPD489 High Dose Range | Placebo
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Change From Baseline in Social Functioning Scale (SFS) at 26 Weeks
Time Frame: Baseline and 26 weeks
Population: Study was discontinued due to non-safety related business prioritization decisions. No subjects were randomized
Arm/Group | SPD489 Low Dose Range | SPD489 High Dose Range | Placebo
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Clinical Global Impression-Schizophrenia Severity of Illness (CGI-SCH-S) Scale
Time Frame: Baseline and week 26
Population: Study was discontinued due to non-safety related business prioritization decisions. No subjects were randomized
Arm/Group | SPD489 Low Dose Range | SPD489 High Dose Range | Placebo
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Clinical Global Impression-Schizophrenia Degree of Change (CGI-SCH-C) Scale
Time Frame: Up to 26 weeks
Population: Study was discontinued due to non-safety related business prioritization decisions. No subjects were randomized
Arm/Group | SPD489 Low Dose Range | SPD489 High Dose Range | Placebo
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Change From Baseline in Amphetamine Cessation Symptom Assessment (ACSA) Total Score at 26 Weeks
Time Frame: Baseline and 26 weeks
Population: Study was discontinued due to non-safety related business prioritization decisions. No subjects were randomized
Arm/Group | SPD489 Low Dose Range | SPD489 High Dose Range | Placebo
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Change From Baseline in Clinical Evaluation of Harmful Behavior (CEHB) Scale at 26 Weeks
Time Frame: Baseline and 26 weeks
Population: Study was discontinued due to non-safety related business prioritization decisions. No subjects were randomized
Arm/Group | SPD489 Low Dose Range | SPD489 High Dose Range | Placebo
Number analyzed (Participants) | 0 | 0 | 0

13. Secondary Outcome: Columbia-Suicide Severity Rating Scale (C-SSRS)
Time Frame: Up to 26 weeks
Population: Study was discontinued due to non-safety related business prioritization decisions. No subjects were randomized
Arm/Group | SPD489 Low Dose Range | SPD489 High Dose Range | Placebo
Number analyzed (Participants) | 0 | 0 | 0

14. Secondary Outcome: Change From Baseline in Calgary Depression Scale for Schizophrenia (CDSS) at 26 Weeks
Time Frame: Baseline and 26 weeks
Population: Study was discontinued due to non-safety related business prioritization decisions. No subjects were randomized
Arm/Group | SPD489 Low Dose Range | SPD489 High Dose Range | Placebo
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Description: Study was discontinued due to non-safety related business prioritization decisions. No subjects were randomized
Arm/Group | SPD489 Low Dose Range | SPD489 High Dose Range | Placebo
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Study was discontinued due to non-safety related business prioritization decisions. No subjects were randomized

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.